CLINICAL TRIAL: NCT05702996
Title: Multicenter, Uncontrolled Pilot Study Evaluating the Efficacy of Eculizumab in the Treatment of Gemcitabine-induced Thrombotic Microangiopathies
Acronym: GEMECULI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/0206/HP
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Thrombotic Microangiopathies
Keywords: Eculizumab; gemcitabine
MeSH Terms: conditions — Thrombotic Microangiopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Thrombotic microangiopathies induced by gemcitabine (Experimental): Patient with Thrombotic microangiopathies induced by gemcitabine will be treat with Eculizumab
  Interventions: Drug: Eculizumab administration

INTERVENTIONS:
Drug: Eculizumab administration — Patient with Thrombotic microangiopathies induced by gemcitabine will be treat with Eculizumab

SUMMARY:
The main objective of this prospective multisite trial is to study the evolution of TMA (thrombotic microangiopathy) induced by gemcitabin and treated by eculizumab.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old 2. Previous treatment with gemcitabine within the last 18 months (duration of treatment ≥ 3 consecutive months and cumulative dose should be ≥ 10 grams). 3. Neoplasia in remission or not in remission but with an estimated life expectancy > 6 months 4. Acute renal failure defined by 1 of the following 2 criteria : Creatinine > 2 times baseline creatinine and/or diuresis < 0.5 ml/kg/h for 12 hours. 5. Clinical and biological criteria for thrombotic microangiopathy: mechanical hemolytic anemia and/or tThrombocytopeniaPatient affiliated with a social security system, 6. Adult patient or representative of the adult patient who has read and understood the information letter and signed the consent form. 7. Woman of childbearing age with effective contraception as defined by the WHO (estrogen-progestin or intrauterine device or tubal ligation) for more than one month and a negative -HCG pregnancy test at baseline, for the duration of the study and for at least 5 months after the end of the treatment, or Postmenopausal woman (non-medically induced amenorrhea for at least 12 months prior to the baseline visit) or For men, use of protection during sexual intercourse for the duration of the study and for at least 60 days after the end of study treatment

Exclusion Criteria:

* 1. Progressive neoplasia with a life expectancy of <6 months 2. Patient with a contraindication to the administration of the treatment experienced: SOLIRIS® 300 mg concentrate for solution for infusion 3. Contraindication to antibiotic prophylaxis 4. Thrombotic microangiopathy associated with cancer (metastatic adenocarcinoma with bone marrow invasion, erythromyelemia, disseminated intravascular coagulation) 5. Active systemic bacterial infection, untreated or confirmed sepsis (positive blood cultures within 7 days of patient inclusion and not treated with effective antibiotic therapy) 6. Unresolved meningococcal infection 7. Patient not vaccinated against meningococcal infection 8. Pregnant or breastfeeding woman or proven lack of contraception 9. Known systemic lupus erythematosus 10. Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection, under guardianship or curatorship 11. Patient participating in another interventional clinical trial / having participated in another interventional clinical trial within 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Time from initiation of eculizumab treatment to renal remission | maximum 12 months

SECONDARY OUTCOMES:
Number of AE and SAE during the study | 12 months
Number of red blood cells transfused before and after treatment with eculizumab | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven GRANGE, MD, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Amiens University Hospital, Amiens
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No